CLINICAL TRIAL: NCT05878392
Title: Comparison Between Different Filling Materials in Immediate Implant
Brief Title: Immediate Implant With Different Filling Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A0103023OS
Record Dates: First submitted 2023-05-09; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Immediate Implant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): immediate implant placement and the buccal jumping gap was packed using PRF
  Interventions: Other: bone filling materials
- group 2 (Experimental): immediate implant placement and the buccal jumping gap was packed using xenograft
  Interventions: Other: bone filling materials
- group 3 (Experimental): immediate implant placement and the buccal jumping gap was packed using alloplast
  Interventions: Other: bone filling materials

INTERVENTIONS:
Other: bone filling materials — the buccal jumping gap was packed using PRF in group 1 the buccal jumping gap was packed using xenograft in group 2 the buccal jumping gap was packed using Alloplastic β-tricalcium phosphate in group 3

SUMMARY:
36 patients, were included in this study. They were chosen from the Outpatient Clinic in the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University for replacement of non-restorable maxillary anterior and premolar teeth (esthetic zone) by immediate implant.

ELIGIBILITY:
Inclusion Criteria:

* Patient medically free from systemic diseases.
* Age above 18 years.
* A single maxillary anterior or premolar tooth that cannot be restored.
* No acute infection is present.
* Patients with sufficient quality and quantity of bone.
* Free from history of bruxism.

Exclusion Criteria:

* A medical condition that would prevent implant surgery.
* Existence of non-treated generalized progressive periodontitis.
* Patients who are smokers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
marginal bone loss | 1 year
  Cone Beam CT (CBCT) was used measure marginal bone loss

SECONDARY OUTCOMES:
Implant Stability: | 1 year
  Resonance frequency analysis (RFA) was used to measure implant stability with an Osstell Mentor device.
Peri-implant Pocket depth | 1 year
  A graduated probe was used to measure the distance between the base of the pocket and the gingival margin

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Elsheikh, Mansoura, Egypt, Egypt

REFERENCES:
- [Derived] Elsheikh HA, Abdelsameaa SE, Elbahnasi AA, Abdel-Rahman FH. Comparison between platelet rich fibrin as space filling material versus xenograft and alloplastic bone grafting materials in immediate implant placement: a randomized clinical trial. BMC Oral Health. 2023 Dec 8;23(1):977. doi: 10.1186/s12903-023-03678-5. PMID 38066454